CLINICAL TRIAL: NCT01742806
Title: Clinical Study for the Impact of Bio-absorbable Felt (NEOVEIL®) With Fibrin Sealant on Removal of Drainage Tube After Minimally Invasive Gastrectomy for Gastric Cancer: Multicenter Prospective Randomized Comparison Study
Brief Title: Clinical Study for the Impact of Bio-absorbable Felt (NEOVEIL®) With Fibrin Sealant on Removal of Drainage Tube After Minimally Invasive Gastrectomy for Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2012-0017
Record Dates: First submitted 2012-11-20; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Minimally invasive surgery; Distal gastrectomy; Bio-absorbable Felt
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): not to use bio-absorbable felt(NEOVEIL®)
- NEOVEIL® (Experimental): To use bio-absorbable felt
  Interventions: Device: bio-absorbable felt(NEOVEIL®)

INTERVENTIONS:
Device: bio-absorbable felt(NEOVEIL®) — To cover bio-absorbable felt over the lymphadenectomy area (hepatoduodenal ligament, #5 and 12/gastroduodenal artery, #6/ pancreas head /suprapancreatic area, #7,8 and 9)
  Other Names: bio-absorbable polyglicolic acid felt,NEOVEIL®
  Arms: NEOVEIL®

SUMMARY:
This study is to evaluate if Bio-absorbable Felt(NEOVEIL®) makes the amount of exudate reduce and shortens time until drain removal after minimally invasive surgery for early gastric cancer.

DETAILED DESCRIPTION:
We investigate the effect on drainage amount of Bio-absorbable Felt(NEOVEIL®) after D1+b or D2 lymphadenectomy with distal gastrectomy for early gastric cancer.

This study is an randomised controlled trial undertaken in 7 centers in South Korea. Patients with stage I-II gastric cancer who is going to have curative distal gastrectomy with D1+b or D2 lymphadenectomy are randomly assigned to use bio-absorbable felt(NEOVEIL®) or not to use it. Block randomisation will be done by a central interactive computerised system, stratified by center.

ELIGIBILITY:
Inclusion Criteria:

* histologic confirmed gastric adenocarcinoma
* Patients who underwent laparoscopic distal gastrectomy.
* preoperative clinical stage I diagnosed with esophagogastroduodenoscopy,endoscopic ultrasonography and computerized tomography.
* patients who underwent more than D1+b lymphadenectomy

Exclusion Criteria:

* Vulnerable participants (pregnant women, under 20 year old, and so on)
* liver or renal disease (Ex. liver cirrhosis, end stage renal disease)
* Transfusion is needed preoperatively or postoperatively due to bleeding
* Preoperative or intraoperative evaluation confirm ascites.
* Patients who use anticoagulant preoperatively or postoperatively

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Time to drain removal | two weeks
  Daily amount of exudate is less than 100cc during consecutive 2 days. There is no evidence of anastomotic leakage, intra-abdominal abscess or bleeding.

SECONDARY OUTCOMES:
total amount of exudate drainage | two weeks
  Total amount of exudate after surgery is recorded.

OTHER OUTCOMES:
Time to discharge after surgery and postoperative complication | up to 30days after randomization
  Time to discharge after surgery and postoperative complication are recorded

CONTACTS AND LOCATIONS:
Overall Officials: WOO JIN HYUNG, M.D. Ph.D., Principal Investigator — Yonsei University
Locations (7):
- South Korea (7):
  - Seoul National University College of Medicine, Bundang Hospital, Seongnam-si, Gyenggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Soonchunhyang University College of Medicine, Bucheon Hospital, Bucheon-si
  - Dong-A University College of Medicine, Busan
  - Seoul National University College of Medicine, Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

REFERENCES:
- [Background] Nakamura T, Shimizu Y, Watanabe S, Hitomi S, Kitano M, Tamada J, Matsunobe S. New bioabsorbable pledgets and non-woven fabrics made from polyglycolide (PGA) for pulmonary surgery: clinical experience. Thorac Cardiovasc Surg. 1990 Apr;38(2):81-5. doi: 10.1055/s-2007-1013999. PMID 2161571
- [Background] Hayashibe A, Sakamoto K, Shinbo M, Makimoto S, Nakamoto T. New method for prevention of bile leakage after hepatic resection. J Surg Oncol. 2006 Jul 1;94(1):57-60. doi: 10.1002/jso.20548. PMID 16788945
- [Background] Ueda K, Tanaka T, Li TS, Tanaka N, Hamano K. Sutureless pneumostasis using bioabsorbable mesh and glue during major lung resection for cancer: who are the best candidates? J Thorac Cardiovasc Surg. 2010 Mar;139(3):600-5. doi: 10.1016/j.jtcvs.2009.06.021. Epub 2009 Aug 4. PMID 19656529